CLINICAL TRIAL: NCT06783686
Title: Effect on Pupil Size After One-time Administration of NV701 (Pilocarpine 1.25%) vs. Vuity (Pilocarpine 1.25%)
Brief Title: Evaluation of NV701 (Pilocarpine 1.25%) Compared With Vuity (Pilocarpine 1.25%) on Pupil Size in Subjects With Presbyopia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Novus Vision LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NV701-02
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pupil Constriction
MeSH Terms: conditions — Miosis | interventions — Pilocarpine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NV701 (Experimental): 1 drop of NV701 (1.25% pilocarpine)
- Vuity (Active Comparator): 1 drop of Vuity (1.25% pilocarpine) in contralateral eye
  Interventions: Drug: Pilocarpine 1.25% Eye drop

INTERVENTIONS:
Drug: NV701 — eye drop
Drug: Pilocarpine 1.25% Eye drop — eye drop
  Arms: Vuity

SUMMARY:
Randomized contralateral eye study to evaluate the effect of one-time dosing of NV701 versus commercially available 1.25% pilocarpine solution on pupil size.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-55 years with presbyopia
* Able to understand and willing to sign the informed consent for the study
* Resting mesopic pupil diameter of >4 mm in both eyes
* Change in mesopic pupil diameter of >1 mm after 1 hour in response to pilocarpine 1.25% in both eyes
* Willing to abstain from contact lens use for 7 days before the study visit
* Women of childbearing age must have a negative urine pregnancy test at the screening visit and be willing to use a reliable method of birth control during the study

Exclusion Criteria:

* Anisocoria >1 mm in photopic or mesopic conditions
* High myopia (-6.00 diopters or greater)
* Any iris abnormality making it difficult to judge pupil diameter as determined by the principal investigator
* Known allergy to any of the study products or medications
* Concurrent use of any topical prescription ophthalmic products
* History of uveitis or intraocular inflammation
* Inability to complete any of the study procedures
* History of ocular surgery other than LASIK or PRK
* History of retinal tear or retinal detachment
* Presence of retinal lattice degeneration, operculated hole, or other retinal pathology on screening exam.
* History of punctal plugs or punctal cautery in one or both eyes
* History of nasolacrimal duct surgery in one or both eyes
* History of blepharoplasty or ptosis surgery in one or both eyes
* History of glaucoma, glaucoma suspect or ocular hypertension diagnosis
* History of acute angle closure or laser peripheral iridotomy
* History of moderate or severe dry eye disease
* Females who are pregnant, nursing, or planning a pregnancy during the study
* Females of childbearing potential and males with partners of childbearing potential who do not agree to use reliable contraception during the study
* Uncontrolled systemic disease

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Change in pupil size over 8 hours | 8 hours
  Area under the curve (AUC) of the change in mesopic pupil diameter over 8 hours after eye drop dosing

SECONDARY OUTCOMES:
Mesopic pupil diameter difference | 8 hours
  Absolute difference in mesopic pupil diameter at 1, 2, 3, 4, 5, 6, 7, and 8 hours after administration

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona Eye Center, Chandler, Arizona
  - Global Research Management, Inc, Glendale, California

IPD SHARING:
Plan to Share IPD: No